CLINICAL TRIAL: NCT00788281
Title: A Multi-Center Randomised Controlled Study to Evaluate Laparoscopic Versus Open Surgery for Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: the department of general surgery, beijing friendship hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJLS01
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy; Conversion to Open Surgery

ARMS (2):
- A (Experimental): laparoscopic surgery plus postsurgery adjuvant chemotherapy of FOLFOX4
  Interventions: Procedure: laparoscopic surgery
- B (Active Comparator): open surgery plus postsurgery adjuvant chemotherapy of FOLFOX4
  Interventions: Procedure: open surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — surgery would be performed by laparoscope
  Arms: A
Procedure: open surgery — surgery would be performed by traditional surgery.
  Arms: B

SUMMARY:
Laparoscopic surgery has been widely accepted for its minimal invasion and safety. However, whether it has the same survival benefit as the traditional open surgery in Chinese population is still unknown. So we designed this study to evaluate the 3 year disease free survival rate in the laparoscopic group versus the open surgery group.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Pathologically confirmed adenocarcinoma
* Pre-surgery image staging as (CT/MRI):T2-3,N0-2,M0,(TNM stage，AJCC，version of 2003)
* Single tumor locating at cecum, ascending colon, descending colon, sigmoid colon, rectosigmoid junction, rectum(distance from anal verge more than 7cm)
* Tumor diameter less than 6cm
* Age 18-75 year
* ECOG 0-2
* Predicted survival longer than 6 months
* Normal liver, renal, bone marrow function: (GPT less than 2 ULN，total bilirubin less than 1.5mg/dl，Cr less than 1.5 ULN，WBC more than 4×109/L，PLT more than 100×109/L)
* No previous history of gastrointestinal surgery
* No previous history of chemotherapy or radiotherapy

Exclusion criteria

* Severe and uncontrolled medical disease including unstable angina pectoris, cardiac infarction and cerebral attack in 6 months
* Could not tolerant general anesthesia or surgery for other organ dis-function
* Allergy to chemotherapeutical agents in the protocol
* History of other malignant tumor within 5 years
* Severe mental disorder
* Continued systematic steroid therapy
* Woman during pregnancy or lactation
* Under study of other clinical trial
* No compliance of the protocol
* Discovery of distant metastasis during surgery
* Postsurgery stage of I or IV tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
disease free survival rate | 3 year
tumor residual rate of LRM and CRM | 1 week
operation mortality | 2 months

SECONDARY OUTCOMES:
survival rate | 3 year
survival rate | 5 year
local recurrence rate | 5 year
operation time | at the end of operation
blood lost | during operation
analgesic dosage | 1,2 and 3 days post surgery
evacuating time | post surgery
operation morbidity | 2 months
transfer to open surgery | during operation
fee | peri-operation

CONTACTS AND LOCATIONS:
Overall Officials: zhongtao zhang, doctor, Principal Investigator — beijing friendship hospital, department of general surgery
Locations (1):
- Beijing Friendship Hospital, Department of General Surgery, Beijing, Beijing Municipality, China